CLINICAL TRIAL: NCT00918034
Title: A Phase 2 Study to Evaluate the Safety and Effectiveness of Using the Litx™ BPH System in Patients With Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH) Who Are Candidates for Interventional Therapy
Brief Title: Study of Light-Activated Talaporfin Sodium in Patients With Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Light Sciences Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSO-OL012
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: BPH; LUTS; talaporfin sodium
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Talaporfin; Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LS11 (talaporfin sodium) (Experimental)
  Interventions: Drug: talaporfin sodium; Device: Transurethral illumination with light emitting diodes; Procedure: Placement

INTERVENTIONS:
Drug: talaporfin sodium — LS11 (talaporfin sodium) dose of 1mg/kg will be administered intravenously by slow push (3-5 minutes)
  Other Names: LS11
Device: Transurethral illumination with light emitting diodes — A light dose of 100 Joules per centimeter (J/cm) will be delivered at 20 mW/cm to each patient for a treatment duration of 1 hour 23 minutes
Procedure: Placement — Placement of device in prostate urethra

SUMMARY:
This is a phase 2 study to evaluate the safety and effectiveness of light-activated talaporfin sodium in patients with LUTS due to benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
This is a phase 2 study to evaluate the safety and effectiveness of using light-activated talaporfin sodium in patients with LUTS due to BPH who are candidates for interventional therapy.

The eligible patient will undergo placement of a proprietary drug activator into the prostatic urethra. Following the placement of the drug activator, patients will receive talaporfin sodium at 1 mg/kg intravenously by slow push over 3-5 minutes. Fifteen minutes after injection a light dose of 100 Joules per centimeter (J/cm) will be delivered at 20 mW/cm to each patient for a treatment duration of 1 hour 23 minutes.

SAE reporting will occur from the day of treatment (Day 0) through end of study (month 12), inclusive. Any SAE that is still ongoing at the end of the study will be followed until assessed as chronic, stable or resolved.

ELIGIBILITY:
Inclusion Criteria:

1. Males, aged 50 years or older with prior diagnosis of BPH;
2. Patients may be eligible whether or not they are on medication for LUTS due to BPH.
3. Patients who are candidates for interventional therapy;
4. Patients who understand and have the ability to sign written informed consent prior to any study procedures and/or discontinuation of exclusionary medications;
5. Patients with an International Prostate Symptom Score of ≥ 15 points;
6. Patients with moderate to severe BPH (Bother Score ≥ 3);
7. Maximum urinary flow rate (Qmax) ≤ 15 mL/sec;
8. Post void residual volume (PVR) ≤ 300 mL;
9. Length of prostatic urethra ≥ 4.0 cm.

Exclusion Criteria:

1. Patients with any previous minimally invasive or surgical intervention for BPH.
2. Patients who are currently enrolled in or who have enrolled in another clinical trial for any disease within the past 30 days.
3. Patients with an active urinary tract infection.
4. Patients with a urethral stricture.
5. Patients with interstitial cystitis.
6. Patients with a predominant middle lobe obstruction.
7. Patients who have evidence or history of prostate or bladder cancer or carcinoma in situ of the bladder.
8. Patients with an abnormal digital rectal exam suggestive of carcinoma of the prostate.
9. Patients with an abnormal digital rectal exam suggestive of an indurated nodule.
10. Patients with a PSA of > 10 ng/ml. If the PSA is 4-10 ng/ml, local standard of care should be pursued to ensure the possibility of prostate cancer is followed up and ruled out prior to, entry into the study.
11. Patients who had a biopsy of the prostate within the past 6 weeks.
12. Patients with bleeding diathesis.
13. Patients with clinically significant renal or hepatic impairment.
14. Patients with neurological conditions felt to affect the bladder or a history of a neurogenic or chronically decompensated bladder.
15. Patients who daily use a pad or device for incontinence.
16. Patients who had an episode of unstable angina pectoris, myocardial infarction, transient ischemic attack, or cerebrovascular accident (stroke) within the past 6 months, or peripheral arterial disease with intermittent claudication or Leriches syndrome.
17. Patient has an interest in future fertility.
18. Patients with prolonged QT interval at baseline and/or who are currently taking medication that prolongs QT interval ("prolonged QT interval" defined as > 450 ms).
19. Inadequate organ function as evidenced by the following: Platelet count <100,000/mm3; WBC <4,000/mm3; Neutrophils <1,800/mm3; Hemoglobin <10 g/dL; AST and ALT >3 x ULN; Creatinine >1.5 x ULN
20. Known sensitivity to porphyrin-type drugs or known history of porphyria.
21. Inability to avoid bright indoor lighting and sunlight during the first 72 hours after LS11 administration.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Safety of light-activated talaporfin sodium by recording of Adverse Events; Preliminary effectiveness of light-activated talaporfin sodium by evaluating the International Prostate Symptom Score (IPSS) along with Bother Score (BS). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sy-Shi Wang, PhD, Study Director — Light Sciences Oncology
Locations (8):
- Australia (3):
  - Royal Brisbane and Women's Hospital Center of Clinical Research, Herston
  - Bayside Urology, Mentone
  - Princess Alexandra Hospital, Wolloongabba
- New Zealand (5):
  - Canterbury Urology Research Trust Hiatt Chambers St. George's Medical Centre, Christchurch
  - Roundhay Medical Centre, Nelson
  - Tauranga Urology Research, Ltd., Tauranga
  - Wellington Urology Research Group Wakefield Urology, Wellington
  - Kensington Hospital Cardinal Points Specialist Centre, Whangarei